CLINICAL TRIAL: NCT03285022
Title: Postoperative Hypersensitivity and Digital Radiographic Assessment of a Zinc Modified Versus a Conventional Glass Ionomer Cement in Deep Carious Lesion: Randomized Controlled Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina mounir elkady, Assisstant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2017-09-17
Record Dates: First submitted 2017-09-14; First posted 2017-09-15 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Carious Dentin
Keywords: Incomplete caries removel; Partial caries removel
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome assessor and participant will be blinded to the type of material
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc modified glass ionomer (Experimental): Zinc modified glass ionomer (chemfill rock) galss ionomer used as restoration for posterior teeth in case of partial caries removel
  Interventions: Procedure: Partial caries removel techniques
- Conventionel glass ionomer (Active Comparator): Conventional glass ionomer used as restoration for posterior teeth in case of partial caries removel
  Interventions: Procedure: Partial caries removel techniques

INTERVENTIONS:
Procedure: Partial caries removel techniques — Removel of all superfacial dentin and leaving the inner affectted dentin
  Other Names: Partial caries removel

SUMMARY:
The study aim to evaluate the difference between the effect of zinc modified glass ionomer and conventional glass ionomer on the success of partial caries removel technique

DETAILED DESCRIPTION:
The zinc ion has an antibacterial effect which could increase the success of partial caries removel technique by decreasing the bactrial population .

ELIGIBILITY:
Inclusion Criteria:

1. Male or female (>18 y)
2. patient with At least 1 deep carious lesion
3. Clinical symptoms of reversible pulpitis with positive pulp response

Exclusion Criteria:

* 1. Patient suffer from irreversible pulpitis (pain with hot or instant pain lasting for a while, resistant to analgesic) 2. Presence of any sign of periapical lesion (like sinus tract ) 3. Teeth with periodontal problem 4. Anterior teeth (material used for non aesthetic region) 5. Pregnant women, to avoid multiple exposure to x ray 6. Patients unable to give consent(mentally retarted, or refuse to right a consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2017-10-20 (Estimated); Primary Completion 2018-04-20 (Estimated); Study Completion 2018-04-20 (Estimated)

PRIMARY OUTCOMES:
Digital radigraphic assessment | At baseline ,3months and 6 months
  The presence of periapical change or change in lamina dura change after the procedure

SECONDARY OUTCOMES:
Post opreative hypersenstivity | Baseline ,at 3 months and at 6 months
  The presence or absence of pain with thermal

IPD SHARING:
Plan to Share IPD: No